CLINICAL TRIAL: NCT05992623
Title: A Pragmatic Randomized Clinical Trial Comparing Rectilinear Biphasic Waveform and Biphasic Truncated Exponential Waveform Shocks for Cardioversion of Atrial Fibrillation (Zoll vs Lifepak)
Brief Title: Clinical Trial Comparing Devices Used for Cardioversion of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U23-04-5042
Record Dates: First submitted 2023-07-21; First posted 2023-08-15 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to a Zoll or Lifepak defibrillator to perform the DCCV. All shocks will be full output (200J for Zoll shocks and 360J for Lifepak shocks). Follow up will be assessment and documentation of rhythm 1 minute after the last shock is delivered. Participants who do not have first shock success will have a second full output shock ≥1 minute after the first shock. Participants who do not have success after a second full output shock will be crossed over to the other defibrillator waveform and receive up to 2 full output shocks with a minimum of 1 minute between each shock to ascertain the outcome of the immediately prior shock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Output synchronized to 200J using Zoll Rectilinear Biphasic Waveform (RBW) defibrillator (Active Comparator): Participants receiving Direct Current Cardioversion (DCCV) using full output Rectilinear Biphasic Waveform (RBW) shocks from a Zoll defibrillator (200 Joules) up to 2 shocks.
  Interventions: Device: Zoll external defibrillator
- Output synchronized to 360J Lifepak Biphasic Truncated Exponential Waveform (BTE) defibrillator (Active Comparator): Participants receiving Direct Current Cardioversion (DCCV) using full output Biphasic Truncated Exponential Waveform (BTE) shocks from a Physiocontrol/Medtronic Lifepak defibrillator (360 Joules) up to 2 shocks.
  Interventions: Device: Lifepak external defibrillator
- Zoll defibrillator waveform used after unsuccessful second full output shock. (Active Comparator): Participants who received first shock via Zoll that do not have success after a second full output shock will be crossed over to the Lifepak defibrillator waveform and receive up to 2 full output shocks with a minimum of 1 minute between each shock to ascertain the outcome of the immediately prior shock.
  Interventions: Device: Lifepak external defibrillator
- Lifepak defibrillator waveform used after unsuccessful second full output shock. (Active Comparator): Participants who received first shock via Lifepak that do not have success after a second full output shock will be crossed over to the Zoll defibrillator waveform and receive up to 2 full output shocks with a minimum of 1 minute between each shock to ascertain the outcome of the immediately prior shock.
  Interventions: Device: Zoll external defibrillator

INTERVENTIONS:
Device: Zoll external defibrillator — Patients with AF will be randomized to receive a full output synchronized 200J shock using a RBW waveform from a Zoll defibrillator
  Arms: Lifepak defibrillator waveform used after unsuccessful second full output shock.; Output synchronized to 200J using Zoll Rectilinear Biphasic Waveform (RBW) defibrillator
Device: Lifepak external defibrillator — Patients with AF will be randomized to receive a full output synchronized 360J shock using a BTE waveform from a Lifepak defibrillator
  Arms: Output synchronized to 360J Lifepak Biphasic Truncated Exponential Waveform (BTE) defibrillator; Zoll defibrillator waveform used after unsuccessful second full output shock.

SUMMARY:
The goal of this single center, investigator initiated, open label prospective randomized controlled trial is to compare the efficacy of a single 200J RBW shock and a single 360J BTE shock. The secondary objective of the study is to compare the frequency of adverse events after one or two 200J RBW or 360J BTE shocks

DETAILED DESCRIPTION:
Data will be derived from approximately 560 patients arriving to Inova sites of care in Atrial Fibrillation (AF) scheduled to undergo either Atrial Fibrillation ablation with expected Direct Current Cardioversion (DCCV) or elective stand-alone AF DCCV. Patients will be included if they are in AF prior to their procedure and are willing to sign the information sheet and comply with the research procedures. Participants will be excluded if they are in a rhythm other than AF on arrival, have not been appropriately anticoagulated with warfarin or direct oral anticoagulant, or have known left atrial appendage thrombus prior to their procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. In AF on presentation with plan for DCCV in either the Electrophysiology lab or DCCV procedure area

Exclusion Criteria:

1. Participants who are receiving any other investigational agents.
2. Parents/guardians or participants who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
3. Patients with arrhythmias other than AF
4. Patients with hemodynamically unstable AF
5. Patients with untreated hyperthyroidism
6. Patients with known or suspected pregnancy
7. Patients without sufficient anticoagulation or a transesophageal echocardiogram or computed tomography scan documenting the absence of intracardiac thrombi

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Atwater, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Health System, Falls Church, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator: Participants receiving Direct Current Cardioversion (DCCV) using full output Rectilinear Biphasic Waveform (RBW) shocks from a Zoll defibrillator (200 Joules) up to 2 shocks.
- 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator: Participants receiving Direct Current Cardioversion (DCCV) using full output Biphasic Truncated Exponential Waveform (BTE) shocks from a Physiocontrol/Medtronic Lifepak defibrillator (360 Joules) up to 2 shocks.
Period: Overall Study
Arm/Group | 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator | 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator
Started | 270 | 276
Completed | 270 | 276
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator | 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator | Total
Number analyzed (Participants) | 270 | 276 | 546
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (13.1) | 68.9 (14.1) | 69.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 90 | 165
  Male | 195 | 186 | 381
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Paroxysmal AF [Number; unit: Participants] | 23 | 31 | 54
Persistent AF [Count of Participants; unit: Participants] | 202 | 193 | 395
Long-standing Persistent AF [Count of Participants; unit: Participants] | 45 | 54 | 99
Prior AF Ablation [Count of Participants; unit: Participants] | 37 | 40 | 77

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants in Normal Sinus Rhythm (NSR) by ECG After the First DCCV Shock
Description: The frequency of NSR by ECG one minute after a single full output DCCV shock is delivered by either a 200J RBW waveform shock from a Zoll Series R defibrillator or 360J BTE waveform shock from a Lifepak 15 defibrillator
Time Frame: At least 1 minute after shock delivery
Measure: Count of Participants; unit: Participants
Groups:
- 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator: Participants receiving Direct Current Cardioversion (DCCV) using full output Rectilinear Biphasic Waveform (RBW) shocks from a Zoll defibrillator (200 Joules)
- 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator: Participants receiving Direct Current Cardioversion (DCCV) using full output Biphasic Truncated Exponential Waveform (BTE) shocks from a Physiocontrol/Medtronic Lifepak defibrillator (360 Joules)
Arm/Group | 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator | 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator
Number analyzed (Participants) | 270 | 276
Participants | 223 | 233
Statistical Analysis 1: Comparison: 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator vs 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator; Test type: Superiority; p = 0.565, Chi-squared

2. Secondary Outcome: The Number of Participants in Normal Sinus Rhythm (NSR) by ECG After the First or Second DCCV Shock
Description: The frequency of NSR by ECG one minute after a first or second full output DCCV shock is delivered using either a 200J RBW waveform shock from a Zoll Series R defibrillator or 360J BTE waveform shock from a Lifepak 15 defibrillator
Time Frame: At least 1 minute after shock delivery
Measure: Count of Participants; unit: Participants
Arm/Group | 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator | 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator
Number analyzed (Participants) | 270 | 276
Participants | 246 | 248
Statistical Analysis 1: Comparison: 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator vs 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator; Test type: Superiority; p = 0.617, Chi-squared

3. Secondary Outcome: The Frequency of NSR One Minute After the First or Second Full Output DCCV Shock is Delivered by a Zoll Series R RBW Waveform Defibrillator and a Lifepak Series 15/20 BTE Waveform Defibrillator After Crossing Over From the Alternative Defibrillator.
Description: The frequency of NSR one minute after the first or second full output DCCV shock is delivered by a Zoll Series R RBW waveform defibrillator and a Lifepak Series 15/20 BTE waveform defibrillator after crossing over from the alternative defibrillator.
Time Frame: At least 1 minute after shock delivery
Population: 24/270 patients failed two consecutive 200J RBW shocks and were eligible for crossover, 2/24 patients exited the protocol prior to crossover. 28/276 patients failed two consecutive 360J shocks from a Lifepak 15 defibrillator and were eligible for crossover, 4/28 patients exited the protocol prior to crossover. Reasons for exiting protocol prematurely included initial conversion followed by reinitiation of AF within 1 minute and intial misinterpretation of atrial flutter as sinus rhythm.
Measure: Count of Participants; unit: Participants
Groups:
- Crossed Over to 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R: Participants receiving Direct Current Cardioversion (DCCV) using full output Rectilinear Biphasic Waveform (RBW) shocks from a Zoll defibrillator (200 Joules) after failing two full output Biphasic Truncated Exponential Waveform (BTE) shocks from a Physiocontrol/Medtronic Lifepak defibrillator (360 Joules)
- Crossed Over to 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak15: Participants receiving Direct Current Cardioversion (DCCV) using full output Biphasic Truncated Exponential Waveform (BTE) shocks from a Physiocontrol/Medtronic Lifepak defibrillator (360 Joules) after failing two full output Rectilinear Biphasic Waveform (RBW) shocks from a Zoll defibrillator (200 Joules).
Arm/Group | Crossed Over to 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R | Crossed Over to 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak15
Number analyzed (Participants) | 24 | 22
Participants | 6 | 12
Statistical Analysis 1: Comparison: Crossed Over to 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R vs Crossed Over to 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak15; Test type: Superiority; p < 0.05, Chi-squared; Mean Difference (Final Values) = 0.04

ADVERSE EVENTS:
Time Frame: 10 minutes
Groups:
- Crossover to 200J RBW Shock After Failed 360J BTE Shock: Participants crossing over to a full output 200J RBW shock from a Zoll defibrillator after 2 failed full output 360J BTE shocks from a Lifepak defibrillator
- Crossover to 360J BTE Shock After Failed 200J RBW Shock: Participants crossing over to a full output 360J BTE shock from a Lifepak defibrillator after 2 failed full output 200J RBW shocks from a Zoll defibrillator
Arm/Group | 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator | 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator | Crossover to 200J RBW Shock After Failed 360J BTE Shock | Crossover to 360J BTE Shock After Failed 200J RBW Shock
All-Cause Mortality (participants affected / at risk) | 0/270 | 0/276 | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/270 | 0/276 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 127/270 | 122/276 | 19/24 | 10/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200J Synchronized Rectilinear Biphasic Waveform (RBW) Shock From Zoll Series R Defibrillator (N=270) | 360J Synchronized Biphasic Truncated Exponential Waveform (BTE) Shock From Lifepak 15 Defibrillator (N=276) | Crossover to 200J RBW Shock After Failed 360J BTE Shock (N=24) | Crossover to 360J BTE Shock After Failed 200J RBW Shock (N=22)
Skin erythema (Skin and subcutaneous tissue disorders) | 115 (115) | 113 (113) | 19 (19) | 9 (9)
Bradycardia/Atriventricular block/ASystole (Cardiac disorders) | 12 (12) | 19 (19) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT05992623/Prot_SAP_000.pdf